CLINICAL TRIAL: NCT00354315
Title: DÉCISION+, a Continuous Professional Development Program to Improve Optimal Drug Prescription : a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Conseil du Médicament du Québec (Unknown)
Responsible Party: France Légaré and Michel Labrecque, Centre hospitalier universitaire de Québec
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CRCHUQ-5-05-12-03; FRSQ-051711
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2008-07

CONDITIONS: Choice Behavior
Keywords: Shared decision making; Optimal drug prescription

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Immediate Continuous medical education (CME)
  Interventions: Behavioral: Continuous medical education (CME)
- 2 (No Intervention): control, 6 months delay CME intervention

INTERVENTIONS:
Behavioral: Continuous medical education (CME) — The intervention will be held over a 6 months period. DECISION+ is a multifaceted intervention program that includes: Interactive workshops (3x180 min), reminders of expected behaviours and feedback.
  Arms: 1

SUMMARY:
The objective of this project is to evaluate the feasibility of a larger randomized trial of the efficacy of DECISION+, a continuous professional development program integrating multiple components, to promote shared decision making concerning drug prescription.

DETAILED DESCRIPTION:
The Conseil du médicament du Québec defines optimal drug use as a "use that maximizes benefits and minimizes risks to population health by taking into account available options, costs and resources as well as patient values and social values". This definition appropriately recognizes the uncertainty surrounding the use of most drugs, i.e. there is often more than one good therapeutic option. The Ottawa Decision Support Framework (ODSF) guides practitioners in assessing decision-making needs in clinical practice, providing support for client decision making, and evaluating the effectiveness of their interventions. DECISION+ is an innovative continuous professional development program for physicians, based on the principles of ODSF and Evidence-Based Medicine. It integrates multiple educational - behavioral change components that aim at promoting optimal shared decision making with respect to drug prescription. The investigators hypothesize that optimal shared decision making should result in optimized prescription behaviors by the physician and optimized drug use by the patient. The objective of this pilot clinical randomized trial of DECISION+ is to evaluate the feasibility of a larger randomized clinical trial, in order to determine the efficacy of the program to promote optimal shared decision making in regards to drug prescription by physicians. This pilot evaluation of the program will focus on one clinical theme: antibiotic prescription for acute respiratory infections (ARI).

The program targets general practitioners and combines three strategies that were proven effective to improve healthcare practices:

1. Interactive workshops
2. Reminders of expected behaviors
3. Feedbacks

Three 180-minute workshops will be held over a six-month period and will include:

1. Retrieval and critical appraisal of information
2. Clinical practice guidelines
3. Acquisition of diagnostic skills
4. Communication of risks and benefits
5. Shared decision making skills
6. Barriers and facilitating factors to optimal shared decision making with respect to drug prescription

Family physicians from four large group practices -the randomization unit- in the province of Québec, Canada will be randomly selected and assigned to one of the following interventions:

1. Immediate DECISION+ antibiotics/ARI program
2. 6-month delayed DECISION+ antibiotics/ARI program

The main outcome measure of this pilot trial is to determine the feasibility of implementing the DECISION+ program on a large scale. Feasibility will be based on the proportion of contacted group practices that agree to participate, the proportion of recruited physicians that participate in the workshops, the level of satisfaction about the workshop, and the proportion of missing data in each survey. Secondary outcomes will include measure of decision to use antibiotics, decisional conflict, decisional regret, prescription profile of antibiotics in ARI, script concordance test, physician' reaction to uncertainty and intention to engage in SDM and to use clinical practice guidelines regarding the use of antibiotics in ARI in future clinical encounters..

The investigators hypothesize that shared decision making will translate into an optimized prescription by the physician and will lead to an optimized drug use by the patient. We believe that this project will help to enhance the health of the Quebec citizen by a better drug use by the patient.

ELIGIBILITY:
Physician: Family medicine group practices (Groupe de médicine familiale) of at least 12 members located in one of the two following regions: Québec and Chaudière-Appalaches, and from which at least 6 members have agreed to participate in the study.

Patients : a) Adult or child consulting a participating physician for an acute respiratory infection (ARI) (i.e. otitis media, rhino-sinusitis, pharyngo-laryngitis, or acute bronchitis), b) Adult or child for whom a treatment with an antibiotic is considered by the patient himself (or guardian, if for a child) or by the physician; c) Patient skills in reading, understanding, and writing French (or guardian, if for a child) equivalent to grade 8; d) Patient (or guardian, if for a child) who can give informed consent for his participation in the study. Patient with a condition requiring emergency care and/or transfer to another care unit will be excluded (e.g.: psychiatric condition, cardiac or pulmonary conditions, a major infection).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
feasibility of a larger RCT aiming at promoting optimal shared decision making in regards to antibiotics prescription by GPs and antibiotics use by patients in acute upper respiratory infections | two years

SECONDARY OUTCOMES:
decision to use antibiotics | one year
decisional conflict | one year
decisional regret | one year
prescription profile of antibiotics in ARI | 18 months
script concordance test | one year
physician' reactions to uncertainty | one year
Intention to engage in SDM and to use clinical practice guidelines regarding the use of antibiotics in ARI in future clinical encounters | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michel Labrecque, MD, Principal Investigator — CHU de Quebec-Universite Laval; France Légaré, MD, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Centre hospitalier universitaire de Québec, Hôpital Saint-François d'Assise, Québec, Quebec, Canada

REFERENCES:
- [Background] Legare F, Labrecque M, Leblanc A, Thivierge R, Godin G, Laurier C, Cote L, O'Connor AM, Allain-Boule N, Rousseau J, Tapp S. Does training family physicians in shared decision making promote optimal use of antibiotics for acute respiratory infections? Study protocol of a pilot clustered randomised controlled trial. BMC Fam Pract. 2007 Nov 29;8:65. doi: 10.1186/1471-2296-8-65. PMID 18047643
- [Derived] Leblanc A, Legare F, Labrecque M, Godin G, Thivierge R, Laurier C, Cote L, O'Connor AM, Rousseau M. Feasibility of a randomised trial of a continuing medical education program in shared decision-making on the use of antibiotics for acute respiratory infections in primary care: the DECISION+ pilot trial. Implement Sci. 2011 Jan 18;6:5. doi: 10.1186/1748-5908-6-5. PMID 21241514
- See also: Study protocol — http://www.biomedcentral.com/1471-2296/8/65/abstract